CLINICAL TRIAL: NCT05023005
Title: Strain-Counterstrain Treatment of Piriformis Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5210286
Record Dates: First submitted 2021-08-11; First posted 2021-08-26 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Low Back Pain, Mechanical; Piriformis Syndrome; Somatic Dysfunction of Sacral Region (Finding)
MeSH Terms: conditions — Low Back Pain; Piriformis Muscle Syndrome; Signs and Symptoms

STUDY DESIGN:
Intervention Model Description: There are two arms to the study: treatment and sham. The treatment group will receive strain-counterstrain for the piriformis muscle. The sham group will receive strain-counterstrain treatment for the hamstring muscle.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant will not know the true positioning for strain counterstrain treatment of piriformis muscle versus hamstring muscle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piriformis Strain-Counterstrain (Experimental): The treatment group will receive strain-counterstrain for the piriformis muscle.
  Interventions: Other: Strain-Counterstrain treatment of piriformis muscle
- Hamstring Strain-Counterstrain (Sham Comparator): The sham group will receive strain-counterstrain treatment for the hamstring muscle.
  Interventions: Other: Strain-Counterstrain treatment of piriformis muscle

INTERVENTIONS:
Other: Strain-Counterstrain treatment of piriformis muscle — Participant will lay prone on table with affected leg close to edge of table. Piriformis muscle tender point is identified and palpated. Then patient leg is passively moved off table and passive hip flexion, abduction, and possible internal/external rotation is added to reduce tender point by 70% or more. This is done passively. This position is held for 90 seconds and then participant is passively returned back to neutral prone position with leg on table. Tender point is palpated again to reassess for change in pain (using subjective visual analog scale). An algometer is also used pre and post to assess objective change in pressure pain threshold.

SUMMARY:
The purpose of this investigator-initiated study is to provide an efficient and non-invasive treatment option for pain caused by the piriformis muscle.

DETAILED DESCRIPTION:
There are two arms to the study: treatment and sham. The treatment group will receive strain-counterstrain for the piriformis muscle. The sham group will receive strain-counterstrain treatment for the hamstring muscle.

There will be two treatments, 1-2 weeks apart ideally.

Participants will fill out the Oswestry Disability Index Questionnaire before the first treatment and after the second treatment (which is 1-2 weeks after the first treatment).

Participants will also identify pain using the Visual Analog Scale (VAS) before and after each treatment. Participants will identify pain at rest prior to treatment using VAS. Participant will then identify pain at the start of treatment while pressure is applied to the piriformis muscle (4.5kg/cm2) and post treatment while pressure is applied to the piriformis muscle (4.5 kg/cm2).

An algometer will be used pre and post each treatment (2 treatments that are 1-2 weeks apart) to objectively measure any change in pain pressure threshold.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* Tender point (or trigger point) in piriformis muscle determined by physical exam

Exclusion criteria:

* Less than 45 degrees of active hip flexion, less than 5 degrees of active hip internal rotation or less than 30 degrees of active hip external rotation, on side of affected piriformis
* Unable to lay prone
* Non-English speaker
* Inability to attend 2 sessions within the same month
* Active cancer
* Pregnant
* Diagnosis of lumbar radiculopathy
* Greater than grade 1 lumbar spondylolisthesis
* Presence of lumbar region Pars Defect
* Receiving massage, acupuncture, chiropractic treatments, osteopathic treatments during study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Algometer - Change in pressure pain threshold | Pre and post each treatment. There are 2 treatments, 1-2 weeks apart from one another.
  Objective improvement in pressure/pain threshold

SECONDARY OUTCOMES:
Change in Visual Analog Scale | Pre and post each treatment. There are 2 treatments, 1-2 weeks apart from one another.
  Subjective improvement in low back/leg pain
Change in Oswestry Disability Index | Before first treatment and after second treatment. Each treatment is 1-2 weeks apart (anticipated).
  Assesses pain with doing different activities (sleeping, walking, sitting, etc), assesses ability to do activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Mickey Lui, Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No